CLINICAL TRIAL: NCT04846777
Title: Brief Smartphone Treatment Study for Anxiety and Depression
Brief Title: Brief Smartphone Treatment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Michelle G. Newman, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00010664
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Generalized Anxiety Disorder
Keywords: Ecological momentary intervention; Mindfulness; Self-help; Digital health; Mobile app
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mindfulness ecological momentary intervention (Experimental): The SMP condition was developed to parallel the treatment while eliminating its theorized active therapeutic elements - open monitoring, acceptance, attending to small moments, breathing retraining, continual practice of mindfulness. Therefore, it did not mention anything about mindfulness at all. Instead, SMP participants were instructed to notice their cognitions and emotions and how distress they might be. No instruction on accepting their thoughts and feelings as they are were given.
  Interventions: Device: Mindfulness ecological momentary intervention
- Self-monitoring placebo (Placebo Comparator): The SMP condition was developed to parallel the treatment while eliminating its theorized active therapeutic elements - open monitoring, acceptance, attending to small moments, breathing retraining, continual practice of mindfulness. Therefore, it did not mention anything about mindfulness at all. Instead, SMP participants were instructed to notice their cognitions and emotions and how distress they might be. No instruction on accepting their thoughts and feelings as they are were given.
  Interventions: Device: Self-monitoring placebo

INTERVENTIONS:
Device: Mindfulness ecological momentary intervention — Access to a smartphone-delivered mindfulness ecological momentary intervention with the Personal Analytics Companion (PACO) app that regularly prompts participants to practice various mindfulness skills at 5 preset times each day.
  Arms: Mindfulness ecological momentary intervention
Device: Self-monitoring placebo — Access to a smartphone-delivered self-monitoring placebo with the PACO app that regularly prompts participants to practice self-monitoring at 5 preset times each day.
  Arms: Self-monitoring placebo

SUMMARY:
Little is known about whether and how brief mindfulness therapies yield clinically beneficial effects. This gap exists despite the rapid growth of smartphone mindfulness applications and presence of mental health treatment gap. Specifically, no prior brief, smartphone mindfulness ecological momentary intervention (MEMI) has targeted generalized anxiety disorder (GAD). Moreover, although theories propose that mindfulness intervention can boost attentional control (AC), executive functioning (EF), perspective-taking, and social cognition skills they have largely gone untested. Thus, this randomized controlled trial (RCT) aims to address these gaps by assessing the efficacy of a 14-day smartphone mindfulness EMI (vs. placebo). Participants with GAD will be randomly assigned to either MEMI or self-monitoring placebo (SMP). Those in treatment will exercise multiple core mindfulness strategies (open monitoring, acceptance, attending to small moments, slowed rhythmic diaphragmatic breathing). Also, those in MEMI will be reminded before bedtime that mindfulness is a lifelong practice. Comparatively, participants assigned to SMP will only be prompted to practice self-monitoring. They will notice their thoughts, rate any distress associated with them, and will not be taught any mindfulness strategies. All prompts will occur 5 times a day, for 14 consecutive days. They will complete self-reports and neuropsychological assessments at pre-, post-, and 1-month follow-up. Multilevel modeling analyses will determine if treatment (vs. self-monitoring placebo (SMP)) produces substantially larger reductions in trait worry and negative perseverative cognitions as well as steeper increases in AC and EF (inhibition, set-shifting, working memory updating). In addition, the investigators hypothesized that MEMI (vs. SMP) would lead to greater increases in performance-based and self-reported trait mindfulness, empathy, and perspective taking. Findings will advance understanding of the efficacy of unguided, technology-assisted, brief mindfulness in a clinical sample.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Generalized Anxiety Disorder based on the Generalized Anxiety Disorder Questionnaire-IV self-report and Mini International Neuropsychiatric Interview
* Current student at the Pennsylvania State University or a community-dwelling adult who expressed interest to participate through the PSU StudyFinder portal
* Expressed interest to seek treatment
* Currently not receiving treatment from a mental health professional
* Able to provide consent
* Proficient in English

Exclusion Criteria:

* Below age 18
* Failure to meet any of above inclusion criteria
* Participant currently undergoing
* Presence of suicidality, mania, psychosis, or substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Generalized Anxiety Disorder Symptoms at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) with categorical ('Yes' for presence and 'No' for absence) and continuous response formats (0 = not at all to 8 = very severely) (Newman et al., 2002) (Item 1 to Item 14 self-report; possible range = 0-12). Generalized Anxiety Disorder Questionnaire-Dimensional (Item 15 to Item 30) with consistent continuous 8-point Likert scale response formats that measures the frequency, intensity, uncontrollability, and degree of excessive worry (e.g., 0 = Always in control to 8 = Never in control) (Newman et al.) (possible range = 0-128). Larger reduction in score denote better outcome.
Change from Baseline Generalized Anxiety Disorder Symptoms at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) with categorical ('Yes' for presence and 'No' for absence) and continuous response formats (0 = not at all to 8 = very severely) (Newman et al., 2002) (Item 1 to Item 14 self-report; possible range = 0-12). Generalized Anxiety Disorder Questionnaire-Dimensional (Item 15 to Item 30) with consistent continuous 8-point Likert scale response formats that measures the frequency, intensity, uncontrollability, and degree of excessive worry (e.g., 0 = Always in control to 8 = Never in control) (Newman et al.) (possible range = 0-128). Larger reduction in score denote better outcome.
Change from Baseline Perseverative Cognitions at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  The 45-item PCQ assessed perseverative cognitive traits linked to anxiety, depressive, and obsessive-compulsive symptoms. Respondents endorsed on a 6-point Likert scale (0 = strongly disagree to 5 = strongly agree). Further, the PCQ-45 comprised six factors: dwelling on the past; expecting the worst; lack of controllability; thoughts discrepant with ideal self; preparing for the future; searching for causes and meanings. Additionally, the PCQ had strong two-week retest reliability, discriminant validity, and convergent validity (Szkodny & Newman, 2019). A total score for PCQ was computed by summing the mean scores from each subscale (total possible score = 0-30). Larger reduction in score denote better outcome.
Change from Baseline Perseverative Cognitions at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  The 45-item PCQ assessed perseverative cognitive traits linked to anxiety, depressive, and obsessive-compulsive symptoms. Respondents endorsed on a 6-point Likert scale (0 = strongly disagree to 5 = strongly agree). Further, the PCQ-45 comprised six factors: dwelling on the past; expecting the worst; lack of controllability; thoughts discrepant with ideal self; preparing for the future; searching for causes and meanings. Additionally, the PCQ had strong two-week retest reliability, discriminant validity, and convergent validity (Szkodny & Newman, 2019). A total score for PCQ was computed by summing the mean scores from each subscale (total possible score = 0-30). Larger reduction in score denote better outcome.

SECONDARY OUTCOMES:
Change from Baseline Depression Symptom Severity at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Beck Depression Inventory (Beck, Steer, & Brown, 1996) (21 of 21 items; self-report; possible range = 0-63). Larger reduction in score denote better outcome.
Change from Baseline Depression Symptom Severity at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Beck Depression Inventory (Beck, Steer, & Brown, 1996) (21 of 21 items; self-report; possible range = 0-63). Larger reduction in score denote better outcome.
Change from Baseline Attentional Control at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Attentional Control Questionnaire (Derryberry & Reed, 2002) (21 of 21 items; self-report; possible range = 0-60). Larger reduction in score denote better outcome.
Change from Baseline Attentional Control at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Attentional Control Questionnaire (Derryberry & Reed, 2002) (21 of 21 items; self-report; possible range = 0-60). Larger reduction in score denote better outcome.
Change from Baseline Working Memory at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV; Wechsler, 2008) (21 of 21 items; self-report; possible range = 0-78). Larger increase in score denote better outcome.
Change from Baseline Working Memory at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV; Wechsler, 2008) (21 of 21 items; self-report; possible range = 0-78). Larger increase in score denote better outcome.
Change from Baseline Set-Shifting at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Trail Making Test Part A and Part B (TMT-A and B; Strauss, Sherman, & Spreen, 2006) (2 of 2 items; self-report; possible range = 0-480). Larger reduction in score denote better outcome.
Change from Baseline Set-Shifting at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Trail Making Test Part A and Part B (TMT-A and B; Strauss, Sherman, & Spreen, 2006) (2 of 2 items; self-report; possible range = 0-480). Larger reduction in score denote better outcome.
Change from Baseline Inhibitory Control at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Color-Word Interference Test response time (Delis, Kaplan, & Kramer, 2001) (1 of 4 items; self-report; possible range = 0-960). Larger reduction in score denote better outcome.
Change from Baseline Inhibitory Control at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Color-Word Interference Test response time (Delis, Kaplan, & Kramer, 2001) (1 of 4 items; self-report; possible range = 0-960). Larger reduction in score denote better outcome.
Change from Baseline Verbal Fluency at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Phonemic cue; category fluency; switching fluency (Delis, Kaplan, & Kramer, 2001) (3 of 3 items; self-report; possible range = 0-240). Larger increase in score denote better outcome.
Change from Baseline Verbal Fluency at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Phonemic cue; category fluency; switching fluency (Delis, Kaplan, & Kramer, 2001) (3 of 3 items; self-report; possible range = 0-240). Larger increase in score denote better outcome.
Change from Baseline Empathy at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Bell-Lysaker Emotion Recognition Test (BLERT; Bryson, Bell, & Lysaker, 1997) (21 of 21 items; self-report; possible range = 0-21). Larger increase in score denote better outcome.
Change from Baseline Empathy at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Bell-Lysaker Emotion Recognition Test (BLERT; Bryson, Bell, & Lysaker, 1997) (21 of 21 items; self-report; possible range = 0-21). Larger increase in score denote better outcome.
Change from Baseline Interpersonal Reactivity Traits at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Interpersonal Reactivity Index (IRI; Davis, 1980) (28 of 28 items; self-report; possible range = 0-140). Larger increase in score denote better outcome.
Change from Baseline Interpersonal Reactivity Traits at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Interpersonal Reactivity Index (IRI; Davis, 1980) (28 of 28 items; self-report; possible range = 0-140). Larger increase in score denote better outcome.
Change from Baseline Trait Mindfulness at 14-Day Post-Treatment | Baseline to 14-Day Post-Treatment
  Five Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2008) (28 of 28 items; self-report; possible range = 0-395). Larger increase in score denote better outcome.
Change from Baseline Trait Mindfulness at 6-Week Post-Randomization | Baseline to 6-Week Post-Randomization
  Five Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2008) (28 of 28 items; self-report; possible range = 0-395). Larger increase in score denote better outcome.

OTHER OUTCOMES:
Mental health disorder screening measures | Baseline
  Generalized anxiety disorder assessed using the Generalized Anxiety Disorder Questionnaire-IV (possible score range = 0 to 14). Higher score indicate worse outcome. Mental health disorders (generalized anxiety disorder, generalized anxiety disorder, major depressive disorder, manic and hypomanic episodes, agoraphobia, panic disorder, post-traumatic stress disorder, alcohol use disorder, substance use disorder, anorexia nervosa, bulimia nervosa, binge eating disorder), as well as rule out organic, drug, or medical causes of mental health problems were determined with the ADIS-5 (Brown & Barlow, 2014). Higher score indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Hani Zainal, M.S., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zainal NH, Newman MG. Who engages? Machine learning insights into digital mindfulness-based intervention for generalized anxiety disorder. J Affect Disord. 2025 Dec 19;399:120963. doi: 10.1016/j.jad.2025.120963. Online ahead of print. PMID 41422949
- [Derived] Zainal NH, Newman MG. Examining the Effects of a Brief, Fully Self-Guided Mindfulness Ecological Momentary Intervention on Empathy and Theory-of-Mind for Generalized Anxiety Disorder: Randomized Controlled Trial. JMIR Ment Health. 2024 May 24;11:e54412. doi: 10.2196/54412. PMID 38787613